CLINICAL TRIAL: NCT05777005
Title: Promoting Smoking Cessation in Campus Via Smoking Cessation Contest: a Chatbot-based Smoking Cessation Intervention
Brief Title: Promoting Smoking Cessation in Campus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Smoking Cessation in Campus
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2023-12

CONDITIONS: Smoking Cessation; Mobile Health
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 5A's/5R's advice+ Chatbot-led group support+ Counselor-led individual support+ health warning leaflet+ Self-help booklet
  Interventions: Behavioral: 5A's/5R's advice; Other: Brief leaflet on health warning and smoking cessation; Other: Self-help smoking cessation booklet; Behavioral: Counselor-led individual support; Behavioral: Chatbot-led group support
- Control group (Active Comparator): 5A's/5R's advice+ Chatbot-led group support+ health warning leaflet+ Self-help booklet
  Interventions: Behavioral: 5A's/5R's advice; Other: Brief leaflet on health warning and smoking cessation; Other: Self-help smoking cessation booklet; Behavioral: Chatbot-led group support

INTERVENTIONS:
Behavioral: 5A's/5R's advice — 5A's (Ask, Advise, Assess, Assist, Arrange) for smokers who are ready to quit, and 5R's (relevance, risks, rewards, roadblocks, and repetition) for smokers who are not ready to quit.
Other: Brief leaflet on health warning and smoking cessation — The contents of the leaflet include the absolute risk of smoking, diseases caused by active and second-hand smoking, horrible pictorial warnings of the health consequences of active and second-hand smoking, and the benefits of quitting.
Other: Self-help smoking cessation booklet — The contents include information about the benefits of quitting, methods to quit, how to handle withdrawal symptoms, misperceptions of quitting, etc.
Behavioral: Counselor-led individual support — Participants will receive three months of counselor-led individual support via WeChat. The regular messages and instant messaging on psychosocial support aim to provide cessation advice, increase self-efficacy and confidence, and social support and behavioral capacity of quitting.
  Arms: Intervention group
Behavioral: Chatbot-led group support — Participants will receive three months of chatbot-led group support via WeChat.

SUMMARY:
This study aims to explore the feasibility, preliminary effectiveness, and implementation outcomes of chatbot-led smoking cessation support in community smokers.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 and above, reside in Zhuhai for the next 6 months;
2. smoke at least 1 cigarette or use e-cigarettes daily;
3. Having a smartphone and a WeChat account, being able to use WeChat skillfully.

Exclusion Criteria:

1. Smokers who have communication barrier (either physically or cognitively);
2. Smokers who are currently participating in other SC programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Participation rate of eligible smokers | Baseline
  the percentage of eligible smokers out of the total number of smokers screened
Biochemical validated quit rate at 6 months follow-up | 6 months follow-up
  The primary outcomes are biochemically validated quit rate (exhaled CO < 4 ppm or salivary cotinine < 30 ng/ml)

SECONDARY OUTCOMES:
Biochemical validated quit rate at 3 months follow-up | 3 months follow-up
  The primary outcomes are biochemically validated quit rate (exhaled CO < 4 ppm or salivary cotinine < 30 ng/ml) at 3-month in the two groups
Self-reported 7-day point prevalence quit rate | 3 and 6 months follow-up
  Self-reported 7-day point prevalence quit rate in the two groups
Smoking reduction rate | 3 and 6 months follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Engagement in chatbot-led group support and/or counselor-led individual support | 3 and 6 months follow-up
  Self-reported engagement in chatbot-led/counselor-led support in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weng X, Yin H, Liu K, Song C, Xie J, Guo N, Wang MP. Chatbot-Led Support Combined With Counselor-Led Support on Smoking Cessation in China: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Sep 23;13:e58636. doi: 10.2196/58636. PMID 39312291